CLINICAL TRIAL: NCT03806439
Title: Post-surgical Delirium in Patients Undergoing Radical Cystectomy.
Status: Not yet recruiting | Type: Observational
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mohammad Hazem I. Ahmad Sabry, Lecturer of Anesthesia, University of Alexandria
Other Study IDs: 16/71(8/2/2017)
Record Dates: First submitted 2019-01-05; First posted 2019-01-16 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Delirium; Radical Cystectomy
MeSH Terms: conditions — Delirium | interventions — Cystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing radical cystectomy.: After approval of local ethical committee and patient consent, the study will be done on patients undergoing radical cystectomy surgery in Alexandria University hospitals from January 5th 2019 till January 4th 2020. The 6-item Cognitive Impairment Test (6CIT) and SPMSQ questionnaire will be used. SPMSQ will be done preoperative and daily for 3 days postoperative, at day 7. Phone call for SPMSQ will be done 3, 6, 9 and 12 months after surgery.
  Interventions: Other: Radical cystectomy.

INTERVENTIONS:
Other: Radical cystectomy. — Adult patients undergoing radical cystectomy.

SUMMARY:
Post-surgical delirium in patients undergoing radical cystectomy. Introduction Delirium occurs after major abdominal surgery may reach about 15% of the patients.(1)

Aim The aim of this study is to determine the incidence of delirium after radical cystectomy surgery and the associated risk factors in Alexandria University hospital.

Patients and Methods After approval of local ethical committee and patient consent, the study will be done on patients undergoing radical cystectomy surgery in Alexandria University hospitals from January 5th 2019 till January 4th 2020. The 6-item Cognitive Impairment Test (6CIT) and SPMSQ questionnaire will be used. SPMSQ will be done preoperative and daily for 3 days postoperative, at day 7. Phone call for SPMSQ will be done 3, 6, 9 and 12 months after surgery.

DETAILED DESCRIPTION:
Post-surgical delirium in patients undergoing radical cystectomy. Introduction Delirium occurs after major abdominal surgery may reach about 15% of the patients.(1)

Aim The aim of this study is to determine the incidence of delirium after radical cystectomy surgery and the associated risk factors in Alexandria University hospital.

Patients and Methods After approval of local ethical committee and patient consent, the study will be done on patients undergoing radical cystectomy surgery in Alexandria University hospitals from January 5th 2019 till January 4th 2020. The 6-item Cognitive Impairment Test (6CIT) and SPMSQ questionnaire will be used. SPMSQ will be done preoperative and daily for 3 days postoperative, at day 7. Phone call for SPMSQ will be done 3, 6, 9 and 12 months after surgery.

Results Results will be collected in tables and graphs. Appropriate statistical analysis will be done.

Discussion Results of the study will be discussed compared to other studies.

ELIGIBILITY:
Inclusion Criteria:Adult patients undergoing radical cystectomy. -

Exclusion Criteria: Patient refusal.

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing radical cystectomy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2028-11-25 (Estimated); Primary Completion 2029-11-24 (Estimated); Study Completion 2029-11-24 (Estimated)

PRIMARY OUTCOMES:
Delirium | 1 year
  Post-surgical delirium in patients undergoing radical cystectomy.

SECONDARY OUTCOMES:
Mortality | 1 year
  Mortality in patients undergoing radical cystectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Hazem I Ahmad Sabry, MB,ChB MD, Principal Investigator — Alexandria University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Raats JW, van Eijsden WA, Crolla RM, Steyerberg EW, van der Laan L. Risk Factors and Outcomes for Postoperative Delirium after Major Surgery in Elderly Patients. PLoS One. 2015 Aug 20;10(8):e0136071. doi: 10.1371/journal.pone.0136071. eCollection 2015. PMID 26291459